CLINICAL TRIAL: NCT05510791
Title: Impact of Nuun SPORT on Subjective Exercise Performance in Male and Female Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Nuun & Company (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of the College of Health Sciences, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PRO-FY2021-417
Record Dates: First submitted 2021-12-08; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Hydration
Keywords: Electrolyte; Running; Nuun

STUDY DESIGN:
Intervention Model Description: randomized, cross-over trial with water control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nuun Sport (Experimental): Citric Acid, Dextrose, Sodium Carbonate, Potassium Bicarbonate, Sodium Bicarbonate, Natural Flavors, Potassium Chloride, Magnesium Oxide, Calcium Carbonate, Stevia Leaf Extract, Avocado Oil, Riboflavin (for color).
  Interventions: Dietary Supplement: Nuun Sport Drink
- Control (Sham Comparator): Water
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Nuun Sport Drink — Subjects will consume a total of 24 ounces water and 1.5 tablets of Nuun SPORT. Specifically, subjects will drink 12 ounces of Nuun drink 15 minutes prior to the 60 min run and 4 ounces of Nuun drink at 15 min, 30 min, and 45 min during the run.
  Arms: Nuun Sport
Dietary Supplement: Control — Subjects will consume a total of 24 ounces water. Specifically, subjects will drink 12 ounces of water 15 minutes prior to the 60 min run and 4 ounces of water at 15 min, 30 min, and 45 min during the run.
  Arms: Control

SUMMARY:
The study will examine the impact of the Nuun Sport tablets, as compared to water only, on heart rate, perceived exertion, and related outcomes in male and female runners, during and following the performance of a 60-minute treadmill run.

DETAILED DESCRIPTION:
As discussed in our prior applications (protocol FY2020-327 and FY2021-96), maintaining adequate hydration is essential to optimal health (Perrier, 2017), as well as athletic performance (Nuccio et al., 2017). When individuals exercise (in particular in a warm environment), they can lose excessive amounts of fluids through sweating, along with necessary electrolytes (e.g., sodium, potassium, chloride). With dehydration, individuals may feel sluggish and can experience impaired physical performance. (Kenefick, 2018)

Many attempts have been made to improve and measure the hydration status of active individuals (Love et al., 2018). This typically involves the ingestion of fluids leading up to activity (typically plain water), as well as the ingestion of fluids during the activity itself (water, along with a diluted carbohydrate/electrolyte beverage).

During aerobic exercise, the shift in fluid (intake versus losses) can affect electrolyte balance, with dehydration and potential adverse effects on performance and health (Perrier et al., 2021; Armstrong et al. 2021). A better understanding of rehydration methods and resultant efficacy would permit selection by an athlete of the optimal method for preventing dehydration to optimize physical performance and reduce potential deleterious effects.

It is well-accepted that electrolyte replenishment is of importance, both during and following exercise-to aid in rehydration for subsequent bouts. Electrolytes (sodium in particular) have been used for decades to aid athlete hydration and this has led to the development of various sport drinks-which also include small amounts of carbohydrate (e.g., Gatorade, Powerade).

The present study will examine the impact of the Nuun Sport tablets, as compared to water only, on heart rate, perceived exertion, and related outcomes: changes in body mass, changes in plasma volume, post-exercise urine volume, and changes in urine specific gravity in male and female runners, during and/or following the performance of a 60-minute treadmill run.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18-29.9 kg/m2 (not obese)
* be able to fast overnight (>8 hrs)
* consuming a minimum of two liters of water per day, on a regular basis
* distance runners: run ≥ 15 miles/week, ≥ 3 runs/week, for at least the past 6 months
* have completed a run of 60 minutes or more at least once per month for the past 6 months
* normal resting blood pressure (systolic < 140 mmHg, diastolic < 90 mmHg) and heart rate (40-80bpm)
* a negative verbal pre-study drug screen (alcohol abuse, amphetamines, benzodiazepines, cocaine, opioids, phencyclidine, barbiturates, cotinine) and no history of use of illicit drugs or other substances of abuse within 12 months of the screening visit

Exclusion Criteria:

* tobacco user
* if female, pregnant
* history of known cardiovascular disease
* more than 400mg caffeine intake per day
* self-reported active infection or illness of any kind
* consumption of alcohol-containing beverages within 48 hours of testing
* consumption of caffeine-containing beverages within 48 hours of testing
* strenuous exercise within 48 hours of testing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Heart rate | baseline
  Heart rate will be measured before and every 10 minutes during the run using a chest strap
Heart rate | 10 minutes into run
  Heart rate will be measured before and every 10 minutes during the run using a chest strap
Heart rate | 20 minutes into run
  Heart rate will be measured before and every 10 minutes during the run using a chest strap
Heart rate | 30 minutes into run
  Heart rate will be measured before and every 10 minutes during the run using a chest strap
Heart rate | 40 minutes into run
  Heart rate will be measured before and every 10 minutes during the run using a chest strap
Heart rate | 50 minutes into run
  Heart rate will be measured before and every 10 minutes during the run using a chest strap
Heart rate | 60 minutes into run
  Heart rate will be measured before and every 10 minutes during the run using a chest strap
Perceived exertion | baseline
  Subjects will self-report perceived exertion using a scale from 0 (no exertion) to 10 (the most exertion)
Perceived exertion | 10 minutes into run
  Subjects will self-report perceived exertion using a scale from 0 (no exertion) to 10 (the most exertion)
Perceived exertion | 20 minutes into run
  Subjects will self-report perceived exertion using a scale from 0 (no exertion) to 10 (the most exertion)
Perceived exertion | 30 minutes into run
  Subjects will self-report perceived exertion using a scale from 0 (no exertion) to 10 (the most exertion)
Perceived exertion | 40 minutes into run
  Subjects will self-report perceived exertion using a scale from 0 (no exertion) to 10 (the most exertion)
Perceived exertion | 50 minutes into run
  Subjects will self-report perceived exertion using a scale from 0 (no exertion) to 10 (the most exertion)
Perceived exertion | 60 minutes into run
  Subjects will self-report perceived exertion using a scale from 0 (no exertion) to 10 (the most exertion)
Specific gravity of urine | baseline
  Specific gravity will be determined from a urine sample
Specific gravity of urine | 15 minutes after run
  Specific gravity will be determined from a urine sample
Plasma Volume | baseline
  Plasma Volume will be determine via blood sampling and determination of hematocrit and hemoglobin
Plasma Volume | 5 minutes after run
  Plasma Volume will be determine via blood sampling and determination of hematocrit and hemoglobin
Body Mass | baseline
  Body Mass will be measured
Body Mass | 5 minutes after run
  Body Mass will be measured
Body Mass | 15 minutes post-run after urine collection
  Body Mass will be measured
Urine output (mass) | 15 minutes post-run
  Urine mass will be determine following collection
Urine output (volume) | 15 minutes post-run
  Urine volume will be determine following collection

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No